CLINICAL TRIAL: NCT04673084
Title: Chest Tube Drainage With Under Water Seal Versus Addition Of Negative Pleural Suction In Chest Trauma Patients
Brief Title: Under Water Seal Versus Negative Pleural Suction in Chest Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yahia Abd almonem Sayed, Chest Tube Drainage With Under Water Seal Versus Addition Of Negative Pleural Suction In Chest Trauma Patients, Assiut University
Other Study IDs: Negative pleural suction
Record Dates: First submitted 2020-10-18; First posted 2020-12-17 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Chest Injury Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: negative pleural suction — by comparing the effect of water seal alone of chest tube in one groups of trauma patients and the effect of both water seal and suction in other group

SUMMARY:
:The investigators aim to provide trauma patient with the best and most efficient managment options and long-term stability with the least complications by comparing the effect of under water seal alone of chest tube in one groups of trauma patients and the effect of both under water seal and suction in other group and the benefits of one versus the other in duration of hospital stay and to assess short-term post-traumatic complications ,also to assess effectiveness of adding suction and patient satisfaction.

DETAILED DESCRIPTION:
Traumas are the leading cause of death in the first four decades of life and are mostly caused by traffic accidents. Thoracic traumas might lead to severe consequences, even though less than 50% of them required a surgical revision. Thoracic traumas can be divided in blunt or penetrating, according to the presence of open wound in the chest. Blunt traumas are the most frequent type of chest trauma with or without rib fractures that might be associated with haemothorax, pneumothorax or haemopneumothorax that are the most typical lesions or laceration.

Pleural chest tubes are used to reestablish negative intrathoracic pressure after disruption of the pleural space. Chest tube positioning is considered necessary in case of a pleural disruption with pneumothorax; intrapleural bleeding causing haemothorax; or in case of pneumo-haemothorax .

The management of pleural chest tubes with primarily under water seal or added suction is the subject of debate, and the benefits of one versus the other in regards to duration of air leak, amount of time the chest tube is in place, length of hospital stay and incidence of complications are unclear.

All of the previous made us interesting to examine the effect of under water seal alone of chest tube in one groups of trauma patients and the effect of both under water seal and suction in other group, the investigators think that power of suction will give the patient better results with less complications and excellent immediate relief with good quality of life, rapid return to normal life .

ELIGIBILITY:
Inclusion Criteria:

* • 1-Pneumothorax after penetrating or blunt chest trauma

  * 2-Hemothorax after penetrating or blunt chest trauma
  * 3-Hemopneumothorax after penetrating or blunt chest trauma 4-All patients of all ages and genders are included

Exclusion Criteria:

* 1-Anyperson associating with body trauma outside chest.

  * 2-Invasive mechanical ventilation
  * 3-Emergent Surgery (thoracoscopy, open thoracotomy)
  * 4-Chronic pulmonary diseases (COPD, CRPD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: : patients who presented to Trauma Department, Assiut University Hospital and who meet the listed inclusion will be eligible for the study. The charts will be reviewed and eligible patients will be filtered.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Decrease duration of hospital stay. | baseline
  We can measure this by:
  Amount and duration of airleak in chest tube.

IPD SHARING:
Plan to Share IPD: No
Overall Goal: We aim to provide trauma patient with the best and most efficient managment options and long-term stability with the least complications by comparing the effect of water seal alone of chest tube in one groups of trauma patients and the effect of both water seal and suction in other group and the benefits of one versus the other in duration of hospital stay and to assess short-term post-traumatic complications ,also to assess effectiveness of adding suction and patient satisfaction.

REFERENCES:
- [Background] Muslim M, Bilal A, Salim M, Khan MA, Baseer A, Ahmed M. Tube thorocostomy: management and outcome in patients with penetrating chest trauma. J Ayub Med Coll Abbottabad. 2008 Oct-Dec;20(4):108-11. PMID 19999219